CLINICAL TRIAL: NCT06880172
Title: Addressing Mental Health and Medication Adherence Among MSM in South Africa
Brief Title: Mental Health and Medication Adherence Among MSM in South Africa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Don Operario, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007894; R34MH135806 (NIH)
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-01

CONDITIONS: HIV
Keywords: MSM; PrEP; ART
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Condition (Experimental): The intervention involves four weekly individual sessions followed by four weekly group support sessions, focusing on themes from the individual sessions. Services will be provided by peer wellness coaches from the MSM community, who will undergo an intensive two-week training with role-play and feedback, followed by weekly supervision. All testing and treatment services are provided free through Aurum.
  Interventions: Behavioral: WeCare
- Control Condition (Active Comparator): The control group (Phase 3) will receive enhanced standard care which includes access to services offered at the POP INN Wellness Clinic including psychoeducation for all individuals who enroll in PrEP or ART services, free medication, enrollment in their standard drop-in Mpowerment support groups, as well as referrals to mental health services on request
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: WeCare — Individual level: Problem identification, Linking Mental health and minority stress, medication adherence, developing an action plan, complementing the plan, and follow-up.
  Group level: Social support and self acceptance in MSM, coping with stigma and minority stress, support for medication adherence
  Arms: Intervention Condition
Behavioral: Standard of Care — Access to services offered at the POP INN Wellness Clinic including psychoeducation for all individuals who enroll in PrEP or ART services, free medication, and enrollment in their standard drop-in. Mpowerment support groups, as well as referrals to mental health services on request
  Arms: Control Condition

SUMMARY:
The goal of this behavioral study is to improve psychological well-being and optimization of HIV prevention and care outcomes for Men who have sex with men (MSM) in South Africa.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) are at an increased risk of HIV infection and transmission, and MSM with depression or anxiety may have adherence to medication challenges. Development of an integrated mental health and adherence support intervention for MSM can be an effective strategy to improve both psychological outcomes and care continuum outcomes including adherence to Pre-Exposure prophylaxis (PrEP) and Anti Retroviral Therapy (ART).

The team proposes developing an intervention approach that responds to the unique social contexts of South African MSM living with or at risk for HIV, and that addresses the relationship between mental health and adherence to HIV prevention medication (daily PrEP) and ART. This intervention approach, WeCare, will adapt an evidence-based program entitled Friendship Bench (i.e., FB) - an empirically supported mental health program using problem-solving therapy (developed/validated in southern Africa) - to incorporate mental health and medication adherence concerns for MSM.

ELIGIBILITY:
Inclusion Criteria:

* Cis-gender male
* Reside in the Johannesburg metropolitan area with no plans to relocate during the next 6 months
* Current prescription for any ART regimen (HIV-positive participants) or daily oral PrEP (HIV-negative participants) at the POP INN clinic
* Self-reported challenges adhering to daily ART (HIV-positive participants) or PrEP (HIV-negative participants)
* Interested in participating in a group discussion to discuss common mental health problems and medication adherence challenges
* Ability to understand and provide informed consent.

Exclusion Criteria:

* Presently engaged in mental health therapy.
* Participated as an intervention participant in a pilot mental health study (AUR6-8-403)
* Refuses audio recording of the focus group discussion
* Those who score over 20 on the PHQ-9 (i.e., indicating severe depression)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cis-gender male (assigned male at birth and identify as male)
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Medication adherence (ART) | Baseline, Month 3, Month 6
  ART adherence will be defined as a suppressed HIV viral load (HIV-1 RNA viral load <200 copies/mL) in the blood sample
Medication adherence (PrEP) | Baseline, Month 3, Month 6
  PrEP adherence is defined as an intracellular TFV-DP concentration ≥700 fmol/punch in a dried blood spot (DBS) sample
Mental health status | Baseline, Month 3, Month 6
  Patient Health Questionnaire (PHQ-9) measures the frequency of depression symptoms within the past two weeks. The PHQ-9 comprises five categories, where a cut-off point of 0-4 indicates no depressive symptoms, 5-9 mild depressive symptoms, 10-14 moderate depressive symptoms, 15-19 moderately-severe depressive symptoms, and 20-27 severe depressive symptoms.
Psychological stress | Baseline, Month 3, Month 6
  The WHO Self-Reporting Questionnaire-20 (SRQ-20) will be used that includes items to reflect symptoms of depression, anxiety and psychosomatic complaints, which are all together grouped under the heading of common mental disorder (CMD).

SECONDARY OUTCOMES:
Status neutral composite adherence | Baseline, Month 3, Month 6
  This is based on TFV-DP concentration ≥700 fmol/punch in a dried blood spot (DBS) sample OR HIV-1 RNA viral load <200 copies/mL)
Self Reported medication adherence | Baseline, Month 3, Month 6
  participants will be asked, "How many days did you not take your PrEP [ART] in the past 30 days (0-30 days)
Persistence | Baseline, 3 months, 6 months
  Defined as time to first PrEP discontinuation, based on a PrEP clinical hold, elective PrEP stop, or missed prescription refill as indicated by pharmacy data

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Pienaar, Principal Investigator — The Aurum Institute, Johannesburg
Locations (1):
- The Aurum Institute, Johannesburg, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Yes
individual participant data that underlie the results reported in this article will be shared after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication (anticipated June 2026)
Access Criteria: Proposals should be directed to don.operario@emory.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third-party website